CLINICAL TRIAL: NCT06314464
Title: Portable Mixed Reality-based Platform for Assessment of Progress in Multisensory Rehabilitation Strategies for Post-TBI Return-to-duty (RTD) Decision Making (Praxis)
Brief Title: Portable Mixed Reality-based Platform for Assessment of Progress in Multisensory Rehabilitation Strategies Post-TBI
Acronym: Praxis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: BlueHalo (Industry)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: C2023.055
Record Dates: First submitted 2024-02-29; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Brain Concussion; Vestibular Disorder; Cognition Disorder; Mild Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Concussion; Dizziness; Vestibular Rehabilitation
MeSH Terms: conditions — Brain Concussion; Vestibular Diseases; Cognition Disorders; Brain Injuries, Traumatic; Dizziness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Praxis (Experimental): Fifteen SMs with post-acute mTBI and residual dizziness/imbalance complaints from the Center for the Intrepid's Special Operations Performance and Recovery (SPaR) Program will receive 4 weeks of Praxis intervention (45 minutes, 5 days per week)
  Interventions: Device: Praxis
- Control (Active Comparator): Fifteen SMs without dizziness/imbalance complaints from the Center for the Intrepid's Special Operations Performance and Recovery (SPaR) Program will receive 4 weeks of supervised cardiovascular activity (45 minutes, 5 days per week)
  Interventions: Behavioral: Supervised cardiovascular exercise

INTERVENTIONS:
Device: Praxis — Praxis' gaze stabilization exercises are delivered via the tablet-based VestAid software that uses the tablet camera to automatically assess compliance in the conduct of vestibulo-ocular reflex exercises. The smooth pursuit, saccade, agility, and dual tasking exercises are delivered in the form of military-themed mixed reality games using the HTC Vive Focus 3 headset.
  Arms: Praxis
Behavioral: Supervised cardiovascular exercise — The supervised cardiovascular exercise does not incorporate gaze stabilization exercises (vestibulo-ocular reflex exercises) or smooth pursuit, saccade, agility, and dual tasking exercises.
  Arms: Control

SUMMARY:
The goal of this comparative pilot study is to provide evidence that Praxis, a portable testbed with low-cost wearable sensors and a mixed reality environment, can deliver effective multisensory rehabilitation exercises with military face-validity in a military service member (SM) population after mild Traumatic Brain Injury (mTBI).

The main questions this comparative pilot study aims to answer are:

* Can the Praxis testbed provide feasible/acceptable 4-week multisensory rehabilitation for SMs with post-acute mTBI?
* Can Praxis detect and influence measurable changes in readiness performance during mTBI recovery?

Fifteen SMs with post-acute mTBI from the Center for the Intrepid's Special Operations Performance and Recovery (SPaR) Program will participate in the multisensory vestibular rehabilitation regimen. These SMs will go through 4 weeks of multisensory vestibular rehabilitation including:

* gaze stabilization
* dual-task balance training
* spatial navigation
* agility training

Data from another fifteen SMs, who will not go through the multisensory rehabilitation regimen and will receive supervised cardiovascular exercise, will be used as the control group.

Researchers will compare the Praxis and Control group to determine if the Praxis group shows improvement over the control group with respect to the military-relevant behavioral performance outcomes and patient-reported symptom scores after the end of the rehabilitation.

DETAILED DESCRIPTION:
This study considers Praxis: a portable testbed with low-cost wearable sensors and a mixed reality environment to deliver effective multisensory rehabilitation exercises with military face-validity. Through a small comparative pilot study, the investigators plan to provide evidence for future multi-center randomized trials (MCRTs) to show that progress in these multisensory exercises correlates with established military readiness assessments; and that the improvements in functional performance in response to multisensory rehabilitation strategies is associated with changes in brain activity.

In preparation for an MCRT, the investigators will conduct a pilot study to examine and settle the issues of feasibility and effectiveness of protocol implementation in accordance with best practices. In this study, we:

* deliver a well-defined rehabilitation strategy via the Praxis system to the enable the patient to practice challenging rehabilitation tasks,
* assess changes in neurophysiological activity via resting state functional magnetic resonance imaging (rs-fMRI) over time in relation to the intensity of the rehabilitation strategy, and
* assess sensitive behavioral outcome measures that monitor the SM's functional gains over time via a battery of military-relevant tasks.

Fifteen SMs with post-acute mTBI from the Center for the Intrepid's Special Operations Performance and Recovery (SPaR) Program will participate in the multisensory vestibular rehabilitation regimen. These SMs will go through 4 weeks of multisensory vestibular rehabilitation:

* gaze stabilization
* dual-task balance training
* spatial navigation
* agility training

Data from another fifteen SMs, who will not go through the multisensory rehabilitation regimen and will receive supervised cardiovascular exercise, will be used as the control group.

The first purposes of this study are to demonstrate the feasibility of obtaining a representative sample of SMs with and without vestibular/ocular impairments post-mTBI in a Special Operations population; determine whether the data is collected reliably; and establish compliance with the protocol in the 4-week study timeline. The primary endpoints for this study are feasibility/acceptability of the 4-week multisensory rehabilitation for SMs with post-acute mTBI as determined by compliance to daily rehabilitation doses as verified by the VestAid software and acceptability measured by the System Usability Scale (SUS) with success thresholds set at 80% or more of the target population completing all the doses and an average total score of 68 or above on the SUS assessment.

The second purpose of this study is to determine the average values and variations of the behavioral outcome measures before and after multisensory rehabilitation delivered by Praxis, as well as the changes in neurophysiological activity, and the correlation between the two. The investigators will use this information to determine the sample size required for a future, larger multicenter study.

The investigators aim to evaluate the effect size relating the implicated functional changes to recovery over the 4-week rehabilitation period in the military population under study. The secondary endpoints of this pilot study will comprise preliminary statistical insights into the ability of Praxis to detect and influence measurable changes in readiness performance during mTBI recovery. The collected metrics include longitudinal Praxis compliance score, pre- and post- behavioral outcome measurements from the readiness battery, and patient-perceived disability questionnaires. Between-group analyses will be conducted to determine the effect size of the Praxis protocol on both the military-relevant behavioral outcomes as well as the patient-reported symptom scores. Within the Praxis group, the investigators will perform an exploratory analysis to examine the correlations between the military-relevant behavioral outcome scores, Praxis compliance scores, and previously implicated objective neurophysiological measures.

ELIGIBILITY:
Inclusion Criteria for Praxis Group:

* Participating in the SPaR Program
* 18-50 years old
* Have a self-reported or clinician-confirmed mTBI
* Have continued complaints of dizziness/imbalance
* Are right-handed as determined by the Edinburgh Handedness Inventory-Short Form

Inclusion Criteria for Control Group:

* Participating in the SPaR Program
* 18-50 years old
* No complaints of dizziness/imbalance

Exclusion Criteria:

* Having impaired mental capacity (e.g., altered capacity due to administration of any mind-altering substances or stress/life situations)
* Displaying behavior that would significantly interfere with validity of data collection or safety during the study
* Reporting significant pain during the evaluation (7/10 by patient subjective report)
* Being pregnant (balance considerations)
* Being unable to abstain from the use of alcohol and medications that might impair participant's balance or cerebral blood flow for 24 hours in advance of testing
* Being mixed or left-handed as determined by the Edinburgh Handedness Inventory-Short Form for the Praxis group undergoing rs-fMRI.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Perceived usability of the Praxis system measured by the System Usability Scale (SUS) | Subjects will be tested after a 4-week intervention period
  The System Usability Scale (SUS) provides an industry-standard reliable tool for measuring the usability of a system (unit of measurement: number, 0-100). This scale relates to the usability (e.g., feasibility) of the prototype device, and is not a health outcome.

SECONDARY OUTCOMES:
Change in Dizziness Handicap Inventory (DHI) score | Subjects will be tested before and after a 4-week intervention period
  The Dizziness Handicap Inventory (DHI) is a 25-item self-assessment inventory designed to evaluate the self-perceived handicapping effects imposed by dizziness (unit of measurement: percentage, 0-100%)
Change in Pittsburgh Sleep Quality Index (PSQI) score | Subjects will be tested before and after a 4-week intervention period
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over the study time interval (unit of measurement: number, 0-21)
Change in Generalized Anxiety Disorder scale (GAD-7) score | Subjects will be tested before and after a 4-week intervention period
  The Generalized Anxiety Disorder scale (GAD-7) is a self-administered patient questionnaire used as a screening tool and severity measure for generalized anxiety disorder (GAD) (unit of measurement: number, 0-21)
Change in Post-Traumatic Stress Disorder Check List - Military Version (PCL-M) score | Subjects will be tested before and after a 4-week intervention period
  The Post-Traumatic Stress Disorder Check List - Military Version (PCL-M) assesses the presence and severity of PTSD symptoms as defined by the Diagnostic and Statistical Manual of Mental Disorders in military personnel (unit of measurement: number, 17-85)
Change in Vestibular Activities Avoidance Instrument-9 (VAAI-9) score | Subjects will be tested before and after a 4-week intervention period
  The Vestibular Activities Avoidance Instrument-9 (VAAI-9) is a patient-reported outcome measure developed to identify fear avoidance beliefs in persons with vestibular disorders (unit of measurement: number, 0-54)
Change in Headache Impact Test-6 (HIT-6) score | Subjects will be tested before and after a 4-week intervention period
  The Headache Impact Test-6 (HIT-6) was developed to measure a wide spectrum of the factors contributing to the burden of headache, and the HIT-6 has demonstrated utility for generating quantitative and pertinent information on the impact of headache. The HIT-6 consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress (unit of measurement: number, 36-78)
Change in Santa Barbara Sense of Direction Scale (SBSOD) score | Subjects will be tested before and after a 4-week intervention period
  The Santa Barbara Sense of Direction Scale (SBSOD) is a standardized self-report scale of environmental spatial ability (unit of measurement: number, 1-7; the average of the 15 items)
Change in time required to perform 300-yard shuttle run (single- and dual-task) | Subjects will be tested before and after a 4-week intervention period
  The 300-yard shuttle run is part of the Ranger Athlete Warrior assessments, and is used to measure anaerobic endurance. The 8-digit grid coordinate memorization task employed in the ReTURN study protocol has been added to provide a cognitive dual-task (unit of measurement: seconds)
Change in perceived fogginess | Subjects will be tested before and after a 4-week intervention period
  Fogginess will be assessed by asking the subject to rate this symptom on a scale from 0 to 10 (as instructed in the Vestibular/Ocular Motor Screening [VOMS], incorporated into the Military Acute Concussion Evaluation 2). (unit of measurement: number, 0-10)
Change in time required to perform 5-10-5 shuttle run | Subjects will be tested before and after a 4-week intervention period
  The 5-10-5 shuttle run is part of the Ranger Athlete Warrior assessments, and is used to measure change in direction / agility. (unit of measurement: seconds)
Change in score for 4-Item Hybrid Assessment of Mobility for mTBI (HAM-4-mTBI) | Subjects will be tested before and after a 4-week intervention period
  The 4-Item Hybrid Assessment of Mobility for mTBI (HAM-4-mTBI) incorporates Functional Gait Assessment's Gait with Horizontal Head Turns and with Pivot Turn, and High Level Mobility Assessment Tool's Fast Forward and Backward Walk (unit of measurement: number, 0-14)
Change in time required to perform POrtable WARrior Test Of Tactical AgiLity (POWAR-TOTAL) (single- and dual-task) | Subjects will be tested before and after a 4-week intervention period
  The POrtable WARrior Test Of Tactical AgiLity (POWAR-TOTAL) is a military-relevant assessment of agility (unit of measurement: seconds)
Change in Vestibular/Ocular Motor Screening (VOMS) total symptom score | Subjects will be tested before and immediately after intervention
  The Vestibular/Ocular Motor Screening (VOMS) total symptom score will be acquired using the Praxis system and include headache, dizziness, nausea, fogginess symptoms scores (unit of measurement: number, 0-40; the sum of the 4 items)
Compliance with 20-minute daily dose of gaze stability exercises | Acquired every 24 hours during the 4-week intervention period
  The compliance with 20-minute daily dose of gaze stability exercises will be acquired using the VestAid system and include the percentage of time (X minutes out of 20 minutes per day) that the subject performed assigned exercises (unit of measurement: percentage, 0-100%)

CONTACTS AND LOCATIONS:
Overall Officials: Pedram Hovareshti, PhD, Principal Investigator — BlueHalo
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hovareshti P, Roeder S, Holt LS, Gao P, Xiao L, Zalkin C, Ou V, Tolani D, Klatt BN, Whitney SL. VestAid: A Tablet-Based Technology for Objective Exercise Monitoring in Vestibular Rehabilitation. Sensors (Basel). 2021 Dec 15;21(24):8388. doi: 10.3390/s21248388. PMID 34960480
- [Background] Hoppes CW, Lambert KH, Whitney SL, Erbele ID, Esquivel CR, Yuan TT. Leveraging Technology for Vestibular Assessment and Rehabilitation in the Operational Environment: A Scoping Review. Bioengineering (Basel). 2024 Jan 25;11(2):117. doi: 10.3390/bioengineering11020117. PMID 38391603
- [Background] Whitney SL, Ou V, Hovareshti P, Costa CM, Cassidy AR, Dunlap PM, Roeder S, Holt L, Tolani D, Klatt BN, Hoppes CW. Utility of VestAid to Detect Eye-Gaze Accuracy in a Participant Exposed to Directed Energy. Mil Med. 2023 Jul 22;188(7-8):e1795-e1801. doi: 10.1093/milmed/usac294. PMID 36208334
- [Derived] Alroumi AM, Hoppes CW, Whitney SL, Li Z, Holt L, Ramakrishnan S, Barnicott SL, Logeais MT, Richard H, Salter SR, Tiede JM, Wirt MD, Hovareshti P. A virtual reality system for delivery of military-specific vestibular rehabilitation after mild traumatic brain injury: the Praxis study protocol. Front Neurol. 2025 May 21;16:1558795. doi: 10.3389/fneur.2025.1558795. eCollection 2025. PMID 40470496